CLINICAL TRIAL: NCT01319955
Title: Influenza Vaccine Efficacy Against Childhood Pneumonia in an Urban Tropical Setting
Brief Title: Flu Vaccine Against Childhood Pneumonia, Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Johns Hopkins University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-09054; 00002579 (Other: Johns Hopkins University)
Record Dates: First submitted 2011-03-09; First posted 2011-03-22 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2016-08

CONDITIONS: Pneumonia; Laboratory Confirmed Influenza
Keywords: Pneumonia; Influenza; Child; Respiratory; Pathogen
MeSH Terms: conditions — Pneumonia; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccine (trivalent inactivated vaccine) (Experimental)
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Inactivated polio vaccine (Active Comparator)
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Two doses of 0.25 ml vaccine delivered IM at least 4 weeks apart.
  Other Names: Vaxigrip Junior

SUMMARY:
Pneumonia is the leading cause of child death worldwide. Data from Bangladesh indicates that influenza has a substantial association with pneumonia among children less than two years old. This study will use commercially available trivalent inactivated vaccine (killed vaccine) to see if it can prevent early childhood pneumonia among children less than two years old. The study will vaccinate children across three seasons (3 years), and look at the effect on the attack rate of pneumonia, as well as its effects on laboratory-confirmed influenza. It will also look at the effect on laboratory-confirmed influenza illness among the non-vaccinated household contacts of all ages of these children.

DETAILED DESCRIPTION:
Pneumonia is the primary cause of child mortality worldwide. The global community is considering interventions to reduce pneumonia burden, including vaccines. Most attention is focused on bacterial vaccines. Influenza vaccine has not received attention due to lack of influenza burden data from high pneumonia endemic settings, and poor understanding of how influenza contributes, independently and with other pathogens, to childhood pneumonia burden. Data from Bangladesh indicate that influenza has a high incidence of over 10% per year among children < 5 years, and that among children who get influenza infection, 28% develop pneumonia, including severe pneumonia. Influenza-infected children who develop pneumonia are significantly younger (< 2y) than those who do not. Due to the high influenza incidence, and the high proportion of influenza-infected children who develop pneumonia, influenza is a major contributor to childhood pneumonia, not only in Bangladesh, but likely throughout the pneumonia endemic tropical and sub-tropical belt. Although trials have been conducted to examine influenza vaccine impact on influenza, none have been conducted specifically to determine the effect on childhood pneumonia, particularly among those < 2 years who are at highest pneumonia risk. We propose to conduct such a trial.

The project goal is to determine whether influenza vaccine (trivalent inactivated vaccine or TIV) can reduce childhood pneumonia burden including: influenza-associated, other aetiology-mediated, and overall pneumonia incidence. The specific objectives are to determine influenza vaccine efficacy on 1) early childhood pneumonia (children < 2 years), 2) laboratory-confirmed influenza and 3) the rates of influenza-specific complications including severe disease, hospitalisation, and otitis media. Secondary objectives include determining the effect of influenza vaccine on household transmission and associated complications among all age groups, the effect on proven non-influenza viral and bacterial invasive diseases, the occurrence of adverse events associated with the vaccine, and to measure immune responsiveness to influenza vaccine in these young children.

Critical milestones include comparison between vaccinated and vaccine-controlled children of 1) pneumonia incidence (vaccine efficacy against pneumonia), 2) influenza incidence (vaccine efficacy against influenza) 3) rates of other clinical syndromes (vaccine efficacy against other childhood morbidity). Milestones related to secondary objectives include comparison between vaccinated and vaccine-controlled children of 1) rates of laboratory-confirmed infection and clinical illness among household contacts and 2) rates of other invasive bacterial and viral diseases, and 3) rates of adverse events. We will also measure childhood immune responsiveness to influenza vaccine and relate that to observed rates of infection and clinical illness.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included if they are de jure residents 6 months to 23 months old at the time of first dose vaccination residing in households under surveillance.

Exclusion Criteria:

* Children will be excluded if they have known chronic respiratory, cardiac, or neurological (including seizure disorders) illnesses, are severely malnourished or require hospitalisation for any other reason, are suspected of having tuberculosis (WHO guidelines) [83], are known to have egg allergy, or parents withhold consent.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3508 (Actual)
Dates: Start 2010-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Clinical pneumonia | Up to 12 months post-vaccination
  Children who present with age-specific tachypnoea, cough with crepitations on auscultation will be determined to have clinical pneumonia. If this occurs ≥14 days post two doses of influenza vaccine, they will be considered fully vaccinated. Comparisons will be made between groups on the number of such episodes.
Laboratory confirmed influenza infection | Up to 12 months post-vaccination
  Influenza infection will be determined by RT-PCR among children with signs and symptoms of febrile and/or respiratory symptoms, including pneumonia.

SECONDARY OUTCOMES:
Indirect effects | Up to 12 months post-vaccination
  Laboratory-confirmed influenza will assessed by RT-PCR among household contacts who present with signs and symptoms of febrile and/or respiratory illness.
Epidemiological and clinical characteristics of influenza infection | Up to 12 months post vaccination
  The epidemiological (seasonality and incidence) and clinical (important clinical syndromes, clinical course, complications and outcomes) characteristics of laboratory-confirmed influenza infection in this age group will be documented.
Effect on non-influenza viral and bacterial invasive disease | Up to 12 months post vaccination
  We will measure the influenza vaccine effect on invasive disease by other pathogens, including pneumococcus, Haemophilus, and several respiratory viruses.
Immunogenicity | Within 4 months of vaccine administration
  We will obtain serum on a 20% subsample of children pre-dose 1, pre-dose 2 and 4 weeks post-dose 2 to determine the immune responsiveness to the vaccine.
Adverse events associated with the vaccine | Beginning Day 0 (day of vaccination) and for the next 7 days
  Adverse events will be monitored, beginning the day of vaccination and for the next 7 days (8 time points) using standardised questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: W. Abdullah Brooks, MD, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Background] Brooks WA, Goswami D, Rahman M, Nahar K, Fry AM, Balish A, Iftekharuddin N, Azim T, Xu X, Klimov A, Bresee J, Bridges C, Luby S. Influenza is a major contributor to childhood pneumonia in a tropical developing country. Pediatr Infect Dis J. 2010 Mar;29(3):216-21. doi: 10.1097/INF.0b013e3181bc23fd. PMID 20190613
- [Derived] Rolfes MA, Goswami D, Sharmeen AT, Yeasmin S, Parvin N, Nahar K, Rahman M, Barends M, Ahmed D, Rahman MZ, Bresee J, Luby S, Moulton LH, Santosham M, Fry AM, Brooks WA. Efficacy of trivalent influenza vaccine against laboratory-confirmed influenza among young children in a randomized trial in Bangladesh. Vaccine. 2017 Dec 15;35(50):6967-6976. doi: 10.1016/j.vaccine.2017.10.074. Epub 2017 Oct 31. PMID 29100706